CLINICAL TRIAL: NCT03726515
Title: Phase 1 Study of EGFRvIII-Directed CAR T Cells Combined With PD-1 Inhibition in Patients With Newly Diagnosed, MGMT-Unmethylated Glioblastoma
Brief Title: CART-EGFRvIII + Pembrolizumab in GBM
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 831706, UPCC 13318
Record Dates: First submitted 2018-10-26; First posted 2018-10-31 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2021-03

CONDITIONS: Glioblastoma
MeSH Terms: conditions — Glioblastoma | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- CART-EGFRvIII + Pembrolizumab (Experimental)
  Interventions: Biological: CART-EGFRvIII T cells; Biological: Pembrolizumab

INTERVENTIONS:
Biological: CART-EGFRvIII T cells — autologous T cells that have been engineered to express an extracellular Humanized single chain antibody (scFv) with specificity for EGFRvIII linked to an intracellular signaling molecule comprised of a tandem signaling domain of the 4-1BB and TCRζ signaling modules.
Biological: Pembrolizumab — humanized monoclonal immunoglobulin (Ig) G4 antibody directed against human cell surface receptor PD-1 (programmed death-1 or programmed cell death-1) with potential immune checkpoint inhibitory and antineoplastic activities.
  Other Names: Keytruda

SUMMARY:
This is an open-label, phase 1 study to assess the safety and tolerability of EGFRvIII T cells in combination with pembrolizumab (PD-1 Inhibitor) in patients with newly diagnosed, EGFRvIII+, MGMT-unmethylated glioblastoma.

ELIGIBILITY:
Inclusion Criteria:

1. One of the following diagnoses of GBM:

   a. Newly diagnosed glioblastoma multiforme that is histologically confirmed by pathology review of surgically resected tissue; OR b. An integrated molecular/pathologic diagnosis of diffuse astrocytic glioma, IDH-wildtype, with molecular features of glioblastoma, WHO grade IV. This diagnosis requires patients have one of the following: i. High-level amplification of EGFR; OR ii. Combined whole chromosome 7 gain and whole chromosome 10 loss (+7/-10); OR iii. TERT promoter mutation.
2. Undergone tumor resection.
3. No prior systemic therapies, radiation, tumor-treating fields, or intratumoral therapeutic agents including Gliadel wafers are allowed. Tumor resection must be the only tumor-directed treatment that the patient has received for glioboblastoma.
4. Tumor tissue is positive for EGFRvIII expression, as performed by either the University of Pennsylvania's in-house fusion transcript panel (RNA-based assay using Illumina HiSeq platform) or NeoGenomics Laboratories (quantitative RT-PCR assay).
5. Tumor tissue is negative for MGMT promoter methylation (i.e. the tumor is MGMT-unmethylated), as performed by either the University of Pennsylvania's in-house pyrosequencing protocol or NeoGenomics Laboratories.
6. Patients ≥ 18 years of age
7. ECOG performance status 0-1
8. Provides written informed consent
9. Must have adequate organ function as measured by:

   1. White blood count ≥ 2500/mm3; platelets ≥ 100,000/mm3, hemoglobin ≥ 9.0 g/dL; without transfusion or growth factor support
   2. AST, ALT, LDH, alkaline phosphatase within 2.5 x upper normal limit, and total bilirubin ≤ 2.0 mg/dL
   3. Serum creatinine < 1.5 x upper limit of normal
   4. Adequate cardiac function (LVEF ≥ 45%)
10. Subjects of reproductive potential must agree to use acceptable birth control methods.

Exclusion Criteria:

1. Pregnant or lactating women
2. Inadequate venous access for or contraindications to leukapheresis.
3. Active Hepatitis B, hepatitis C, or HIV infection, or other active, uncontrolled infection
4. History of allergy or hypersensitivity to study product excipients (human serum albumin, DMSO, and Dextran 40)
5. History of severe hypersensitivity reactions to other monoclonal antibodies which in the opinion of the investigator may post an increased risk of serious infusion reactions.
6. Requirement for immunosuppressive agents including but not limited to cyclosporine, MMF, tacrolimus, rapamycin, or anti-TNF agents within 4 weeks of eligibility confirmation by the physician-investigator.
7. Subjects with a history of known or suspected, severe or uncontrolled autoimmune or connective tissue disease. Patients with vitiligo, controlled type 1 diabetes mellitus (on stable insulin dose), residual autoimmune-related hypothyroidism (due to autoimmune condition only requiring hormone replacement), or psoriasis (not requiring systemic treatment), or conditions not expected to recur in the absence of an external trigger, are permitted to enroll.
8. Known history or current interstitial lung disease or non-infectious pneumonitis
9. Prior allogenic bone marrow or solid organ transplant

11. Any uncontrolled active medical or psychiatric disorder that would preclude participation as outlined.

12. Severe, active co-morbidity in the opinion of the physician-investigator would preclude participation in this study, including but not limited to the following:

1. Unstable angina within 6 months prior to eligibility confirmation by the physician-investigator
2. Transmural myocardial infarction within the last 6 months prior to eligibility confirmation by the physician-investigator
3. New York Heart Association grade II or greater congestive heart failure requiring hospitalization within 12 months prior to eligibility confirmation by the physician-investigator.
4. Serious and inadequately controlled cardiac arrhythmia
5. Serious or non-healing wound, ulcer, or history of abdominal fistula, gastrointestinal perforation, intra-abdominal abscess major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to eligibility confirmation by the physician-investigator, with the exception of the craniotomy for tumor resection.

   13. Patients with tumors primarily localized to the brain stem or spinal cord.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2019-03-11 (Actual); Primary Completion 2021-02-27 (Actual); Study Completion 2021-02-27 (Actual)

PRIMARY OUTCOMES:
Number of subjects with treatment-related adverse events, using NCI CTCAE v5.0. | 15 Years

SECONDARY OUTCOMES:
Overall survival Rate | 15 Years
  Number of days from the date of the first CART-EGFRvIII infusion to the date of death of any cause. The survival function of OS will be calculated by the Kaplan-Meier method.
Progression-free survival (PFS) | 15 Years
  The number of days from the date of the first CART-EGFRvIII infusion to the first documented disease progression (based on standard MRI evaluation using the modified RANO criteria) or date of death, whichever occurs first. PFS will be calculated by the Kaplan-Meier method.
Objective response rate (ORR) | 15 Years
  The proportion of patients with complete response (CR) or partial response (PR) out of the total number of efficacy evaluable subjects. Exact 90%confidence interval for ORR will be computed.

CONTACTS AND LOCATIONS:
Overall Officials: Donald O'Rourke, MD, Principal Investigator — Abramson Cancer Center at Penn Medicine
Locations (1):
- Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania, United States